CLINICAL TRIAL: NCT00707824
Title: Study of Epidural Nalbuphine for Prevention of Epidural Morphine Induced Pruritus
Brief Title: Epidural Nalbuphine for Postcesarean Epidural Morphine Induced Pruritus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Assistant Professor Orawan Pongraweewan, Mahidol University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 110/2000
Record Dates: First submitted 2008-06-29; First posted 2008-07-01 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2006-02

CONDITIONS: Cesarean Section
Keywords: pruritus; epidural morphine
MeSH Terms: conditions — Pruritus | interventions — Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): 1= placebo
  Interventions: Other: NSS
- 2 (Active Comparator): 2=nalbuphine 5 mg
  Interventions: Drug: nalbuphine
- 3 (Active Comparator): 3=nalbuphine 10 mg
  Interventions: Drug: nalbuphine

INTERVENTIONS:
Drug: nalbuphine — nalbuphine 5 mg epidural
  Other Names: nubain
  Arms: 2
Drug: nalbuphine — nalbuphine 10 mg epidural
  Other Names: nubaine
  Arms: 3
Other: NSS — NSS
  Other Names: nornal saline
  Arms: 1

SUMMARY:
Can epidural nalbuphine reduce incidence or severity of epidural morphine induced pruritus in patient undergoing cesarean section?

DETAILED DESCRIPTION:
182 parturients,ASA 1-2 undergoing cesarean section under epidural block were enrolled in the study. After obtaining informed consent,all received epidural anesthesia using 2% lidocaine with epinephrine 1:200000 via epidural cathetes at L2-3 or L3-4 in a volume suffient to achieve a T4 sensory level bilaterally.

After the umbilical cord was clamped,patients were assigned randomly to three groups.The placebo group,N-5 group,and N-10 group received 4 ml epidural solution containing morphine 4 mg plus either saline, nalbuphine 5 mg, and nalbuphine 10 mg respectively.At the post anesthetic care unit, intravenous pethidine PCA were administered for inadequate pain control.

Outcome measures :

Incidence and severity of postoperative pruritus Quality of pain control Side effects of epidural morphine and nalbuphine such as respiratory depression,sedation

ELIGIBILITY:
Inclusion Criteria:

* full term parturient undergoing elective cesarean section
* ASA 1-2

Exclusion Criteria:

* drug or alcohol abuses
* contraindication for regional anesthesia
* received opioids within 12 hours

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2000-06; Primary Completion 2005-12 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
incidence and severity of pruritus | 24 hr

SECONDARY OUTCOMES:
visual analogue pain score | 24 hr

CONTACTS AND LOCATIONS:
Overall Officials: Orawan Pongraweewan, MD, Principal Investigator — Mahidol University
Locations (1):
- Mahidol University, Bangkoknoi, Bangkok, Thailand